CLINICAL TRIAL: NCT02918487
Title: Role of Breathe Free® in the Management of Bronchial Asthma- A Randomized Placebo Controlled Trial
Brief Title: Role of Herbs in the Management of Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OI - 004 - 2016
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): [Formoterol + Fluticasone] Single maintenance and reliever therapy(SMART) and Active polyherbal capsule
  Interventions: Drug: Polyherbal; Drug: Placebo
- Placebo (Placebo Comparator): [Formoterol + Fluticasone] conventional along with inert similar looking placebo capsules
  Interventions: Drug: Polyherbal; Drug: Placebo

INTERVENTIONS:
Drug: Polyherbal — Each capsule contains four herbs: Inula racemosa, Ocimum sanctum, Terminalia Belerica and Piperum longum
  Other Names: Breathe Free
Drug: Placebo — Inactive compound that is similar looking as the intervention

SUMMARY:
The aim of this trial is to study the effect of a polyherbal capsule containing four herbs: Inula racemosa, Ocimum sanctum, Terminalia Belerica and Piperum longum in the treatment of bronchial asthma.

DETAILED DESCRIPTION:
A randomized placebo controlled double blind trial. Four herbs that have proven efficacy on bronchial asthma will be given. Equally matched placebo will be given randomly to patients. Each arm active herbs and placebo will be compared against the Formoterol+Fluticasone Single maintenance and reliever therapy(SMART) and conventional therapy. All the parameters of Bronchial Asthma(BA) will be compared between the randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years.
* History of asthma documented by a physician for at least 6 months
* Patients on steroid therapy for at least 4 weeks.
* If not on steroid therapy, patient and physician must be willing for 4 weeks run in on steroid therapy.
* The subject agrees to participate in the study

Exclusion Criteria:

* Any one of the following

  * Acute illness (such as cold, flu, etc.) within one week before the administration of study drug
  * Abnormal hepatic and renal function
  * Pregnant, attempting to conceive, or lactating women
  * Current or former employees of organic India
  * Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.
  * Physician uncomfortable with patient compliance to treatments or follow up.
  * Non-compliance to tobacco cessation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with 15% increase in forced expiratory volume(FEV1) from baseline | 6 months
Number of patients with 50 L/min peak expiratory flow rate(PEFR) from baseline | 6 months

SECONDARY OUTCOMES:
Number of patients with frequency of asthma exacerbation per week | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alben Sigamani, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Mazumdar Shaw Mutispeciality Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided